CLINICAL TRIAL: NCT02426411
Title: A Double-blind, Placebo-controlled, Randomized Dose Ranging Trial to Determine the Safety and Efficacy of Two Dose Levels of EMA401 in Patients With Postherpetic Neuralgia
Brief Title: Dose Ranging Trial to Determine the Safety and Efficacy of EMA401 in Patients With PHN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Spinifex Pharmaceuticals Pty Ltd (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMA401-006
Record Dates: First submitted 2015-04-17; First posted 2015-04-24 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — EMA400

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- EMA401 200 mg (Experimental): 2 X 50 mg capsules BID
  Interventions: Drug: EMA401 200 mg
- EMA401 600 mg (Experimental): 2 X 150 mg capsules BID
  Interventions: Drug: EMA401 600 mg
- Placebo (Placebo Comparator): Placebo to match 2 capsules BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EMA401 200 mg
  Arms: EMA401 200 mg
Drug: EMA401 600 mg
  Arms: EMA401 600 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study is a randomized, double blind, placebo-controlled, parallel-group comparison (two dose levels of EMA401 versus a placebo group), of safety and efficacy in patients with postherpetic neuralgia.

DETAILED DESCRIPTION:
Screening Period (Up to Four Weeks) to confirm eligibility for the study which will be determined by Screening tests, physical examination/medical history and fulfillment of eligibility criteria including assessment of pain.

Study Period (14 Weeks) Approximately 360 eligible male and female patients will receive double-blind treatment for 14 weeks. Patients will be randomized in a 1:1:1 ratio to treatment with EMA401 100 mg BID, 300 mg BID or placebo.

Patients will attend the study site at the end of the Baseline visit and end of Weeks 1, 3, 5, 7, 9, 11, 13, and 14 for on-study assessments.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed as suffering from PHN defined as pain in the region of the rash persisting for more than six months after onset of herpes zoster rash.
* Be assessed as suffering from moderate to severe pain across the Screening Period. The assessment of moderate and severe pain will be made using an algorithm proprietary to Spinifex. The Investigator/site staff will be informed immediately as to whether the patient is eligible or ineligible on the ePRO website based on the patient entering all relevant pain scores in the eDiary device.
* Women of child bearing potential (WOCBP) must have a negative urine pregnancy test at the Screening Visit (Visit 1) and within 72 hours prior to administration of IP.

Exclusion Criteria:

* Patients taking any topical treatment for their PHN at the time of Screening Visit 2 will be excluded, including lidocaine plaster, capsaicin patch, and any other topical preparations of these or any other topical medications (e.g., aspirin, Non-Steroidal Anti-Inflammatory Drugs (NSAIDs)) for their PHN.
* Have a blood pressure reading, after resting for at least five minutes, outside a systolic blood pressure range of 84-151 mmHg or a diastolic blood pressure > 95 mmHg. If the blood pressure is outside of the range, a repeat measurement can be taken after the patient has rested. The repeat measurement should be used as the screening value.
* Have serum aspartate transaminase (AST) or alanine transaminase (ALT) levels > 1.5 x the upper limit of normal or have total bilirubin concentrations > 1.5 x the upper limit of normal at Screening (Visit 1).
* Patients who have a known diagnosis of diabetes and are stable on medication with a hemoglobin A1c > 8%. Those who do not have a known diagnosis of diabetes with a hemoglobin A1c > 7%.
* Have active herpes zoster upon physical examination at Screening (Visit 1) or during the study.
* Known history of, or positive laboratory result for hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection as defined by being seropositive for hepatitis B surface antigen (HBsAg), HCV antibodies or HIV antibodies respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of two dose levels of EMA401 compared to placebo in patients with postherpetic neuralgia (PHN), as assessed by the change in the weekly mean of the 24 hour average pain score using an 11-point Numerical Rating Scale (NRS) | Baseline to approximately Week 14

SECONDARY OUTCOMES:
To evaluate the effect of EMA401 compared to placebo on the Brief Pain Inventory-Short Form (BPI-SF) interference total score | Baseline to approximately Week 14
To evaluate the effect of EMA401 compared to placebo on the weekly mean of the 24 hour worst NRS pain score | Baseline to approximately Week 14
To evaluate the effect of EMA401 compared to placebo on the Patient Global Impression of Change (PGIC) | Baseline to approximately Week 14
To evaluate the effect of EMA401 compared to placebo on the BPI-SF average pain | Baseline to approximately Week 14
To determine the proportion of EMA401 patients achieving a ≥ 30% and a ≥ 50% reduction in weekly mean pain of the 24 hour average score (NRS) compared to placebo (i.e., responder rates) | Baseline to approximately Week 14
To evaluate the effect of EMA401 compared to placebo on the Insomnia Severity Index (ISI) | Baseline to approximately Week 14
To evaluate the safety and tolerability of EMA401 in patients with PHN as measured by adverse events, vital signs, and laboratory results | Baseline to approximately Week 14